CLINICAL TRIAL: NCT03747809
Title: Cost-effectiveness Analysis on Remote Monitoring for Cardiovascular Electronic Implantable Devices in Japan by Using Systematic Review Methodology - 2018 Reimbursement Update
Brief Title: Cost-effectiveness Analysis on Remote Monitoring for CIEDs in Japan by Using Systematic Review Methodology
Status: Completed | Type: Observational
Sponsor: The Open University of Japan (Other)
Responsible Party: Principal Investigator, Tomoya SHIRANE, Principal Investigator, The Open University of Japan
Other Study IDs: OUJ11200212018111801
Record Dates: First submitted 2018-11-17; First posted 2018-11-20 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Cardiovascular Diseases; Heart Failure
Keywords: Remote Monitoring
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Patients with CIEDs having Remote Monitoring
  Interventions: Device: CIEDs Remote Monitoring System
- Patients with CIEDs having no Remote Monitoring

INTERVENTIONS:
Device: CIEDs Remote Monitoring System — Cardiac device remote monitoring system
  Groups: Patients with CIEDs having Remote Monitoring

SUMMARY:
2018 Revision of Health Reimbursement in Japan recognized non face-to-face diagnostics, such as Online Treatment, as the standard of care. There was a significantly additional cost for Cardiovascular Implantable Electronic Devices (CIEDs) Management Fee as well. The adaption of Remote Monitoring for CIEDs patients is recommended by the societies based on the clinical evidences. However, how QALYs earned by CIEDs Remote Monitoring are justified in Japanese reimbursement environment from the cost-effectiveness standpoint is still not so clear. The evaluation about the impact on the health economics about the installation of CIEDs Remote Monitoring has not been enough due to the lack of the researches around this field. Therefore this research is designed to examine the impact of the installation of CIEDs Remote Monitoring from the health economics perspective by considering the health insurance system and the clinical process in Japan, through Systematic Review methodology.

DETAILED DESCRIPTION:
2018 Revision of Health Reimbursement in Japan recognized non face-to-face diagnostics, such as Online Treatment, as the standard of care. There was a significantly additional cost for Cardiovascular Implantable Electronic Devices (CIEDs) Management Fee as well. The adaption of Remote Monitoring for CIEDs patients is recommended by the societies based on the clinical evidences. However, how QALYs earned by CIEDs Remote Monitoring are justified in Japanese reimbursement environment from the cost-effectiveness standpoint is still not so clear. The evaluation about the impact on the health economics about the installation of CIEDs Remote Monitoring has not been enough due to the lack of the researches around this field. Therefore this research is designed to examine the impact of the installation of CIEDs Remote Monitoring from the health economics perspective by considering the health insurance system and the clinical process in Japan, through Systematic Review methodology.

ELIGIBILITY:
Inclusion Criteria:

* Studies that involves CIEDs Remote Monitoring, such as Implantable Cardioverter Defibrillator, Cardiac Resynchronization Therapy, and Pacemaker
* Follow-up periods more than or equal to 12 months
* Prospective studies
* QALYs available to make ICER analysis possible
* Published after Year of 1971

Exclusion Criteria:

* Studies that are not related with CIEDs
* Follow-up periods less than 12 months
* Not prospective studies
* QALYs unavailable
* Published before Year or 1971

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults implanted with CIEDs such as Implantable Cardioverter Defibrillator, Cardiac Resynchronization Therapy, or Pacemaker
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-16 (Actual); Study Completion 2019-06-16 (Actual)

PRIMARY OUTCOMES:
Differences of ICERs based on earned QALYs from selected studies by applying to Japanese reimbursement environment. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Open University of Japan, Chiba, Japan

IPD SHARING:
Plan to Share IPD: Undecided